CLINICAL TRIAL: NCT05236699
Title: Single-arm, Multicenter II Phase Clinical Study of DEB-TACE Combined With Surufatinib and Camrelizumab in the Treatment of Inoperable or Metastatic Intrahepatic Cholangiocarcinoma
Brief Title: A Clinical Study of DEB-TACE Combined With Surufatinib and Camrelizumab in the Treatment of Inoperable or Metastatic ICC
Acronym: CCGLC-005
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Wan-Guang Zhang, Prof., Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-SPRING-B105
Record Dates: First submitted 2021-10-24; First posted 2022-02-11 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: DEB-TACE; Surufatinib; Camrelizumab
MeSH Terms: conditions — Cholangiocarcinoma | interventions — surufatinib; camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DEB-TACE combined with Surufatinib and Camrelizumab (Experimental)
  Interventions: Combination Product: DEB-TACE combined with Surufatinib and Camrelizumab

INTERVENTIONS:
Combination Product: DEB-TACE combined with Surufatinib and Camrelizumab — 1. All patients will be treated with standard DEB-TACE on the first day (D1).
  2. After DEB-TACE, if the liver function is Child-PughA grade, they will be treated with Camrelizumab on the same day, 200mg/ times, intravenous injection, once every 3 weeks.
  3. Surufatinib capsule will be given orally to 250mg within 1 hour after breakfast on the second day (D2) after the first DEB-TACE. The drug will be given continuously once a day and stopped on the same day of each DEB-TACE.
  4. The combination of drugs for 3 weeks is a cycle.The treatment will continue until the patient developed the disease or met the other criteria for terminating the study.

SUMMARY:
At present, for advanced Intrahepatic Cholangiocarcinoma（ICC）, the effect of single treatment is not good.So far, superselective drug-eluting bead transarterial chemoembolization（DEB-TACE） is a good method for the treatment of local lesions in advanced ICC.Studies have shown that the combination of sovantinib and immunotherapy has also shown encouraging results, and patients are well tolerated.Therefore, we designed DEB-TACE combined with Surufatinib and Camrelizumab for the exploratory study of inoperable or metastatic ICC, in order to provide a safe, effective and tolerable option for patients with ICC, prolong their survival time and improve their quality of life.

DETAILED DESCRIPTION:
Study design:

This is a single-arm, open, multicenter II phase clinical study to compare the efficacy and safety of DEB-TACE combined with Surufatinib and Camrelizumab in the treatment of inoperable or metastatic ICC.

Study population:

20 untreated patients with inoperable or metastatic intrahepatic cholangiocarcinoma

Treatment:

1. All patients were treated with standard DEB-TACE on the first day (D1).
2. Immediately after the first DEB-TACE, the liver function was reexamined. If the liver function was grade Child-Pugh A, Camrelizumab was given intravenously once every 3 weeks (D1) on the same day, 200mg/, once every 3 weeks (D1).
3. Surufatinib capsule was given orally to 250mg within 1 hour after breakfast on the second day (D2) after the first DEB-TACE. The drug was given continuously once a day and stopped on the same day of each DEB-TACE.
4. The combination of drugs for 3 weeks is a cycle.The treatment continued until the patient developed the disease or met the other criteria for terminating the study.

Curative effect evaluation： The tumor condition was evaluated by imaging method at D28 (±7 days) after each DEB-TACE, until the curative effect was evaluated as PD or unsuitable for further treatment. After 3 times of DEB-TACE treatment, the tumor efficacy was evaluated every 12 weeks (±7 days) from 6 months after the first DEB-TACE treatment until disease progression (Response Evaluation Criteria In Solid Tumors（RECIST）1.1) or death (during treatment) or toxicity intolerable. The tumor treatment and survival status after disease progression were recorded.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily joined the study and signed an informed consent form with good compliance and follow-up.
* Inoperable or metastatic intrahepatic cholangiocarcinoma diagnosed by histopathology or cytology;
* In accordance with the diagnostic criteria of NCCN guidelines for intrahepatic cholangiocarcinoma, the diagnosis of intrahepatic cholangiocarcinoma that is not suitable for radical resection: unable to obtain R0 resection, multiple liver, lymph node metastasis beyond the hilar area and distant metastasis;
* ECOG score: 0-1; expected survival ≥ 12 weeks;
* Liver function Child-Pugh A grade
* Patients who have not received systematic treatment for unresectable or metastatic biliary tract cancer; those who have received adjuvant or neoadjuvant chemotherapy and relapse 6 months after the end of chemotherapy can be enrolled in the group.
* At least one measurable lesion (according to RECIST1.1 standard); its diameter ≥ 1cm was accurately measured by magnetic resonance imaging (MRI) enhancement or computed tomography (CT) enhancement, and the target lesion had not received local treatment in the past (including not limited to hepatic arterial Infusion chemotherapy, radiofrequency ablation, argon-helium knife, radiotherapy, etc.);
* No serious organic diseases of heart, lung, brain and other organs;
* The functions of major organs and bone marrow are basically normal:

  1. Blood routine: WBC ≥ 4.0x10^9/L, neutrophils ≥ 1.5x10^9/L, platelets ≥ 80x10^9/L, hemoglobin ≥ 90 g/L
  2. International standardized ratio (INR) ≤ 1.5 × upper limit of normal value (ULN), and activated partial thromboplastin time (APTT) ≤ 6sbot
  3. liver function: serum total bilirubin ≤ 2xULN ;ALT/ AST ≤ 2xULN; serum albumin ≥ 28g/L.
  4. Renal function: serum creatinine ≤ 1.5xULN or eGFR ≥ 60%, and creatinine clearance rate (CCr) 60ml / min; excluding urinary tract infection, urine routine showed that urinary protein < 2+, 24-hour urine protein should be collected from ≥ 2 + patients < 1g
  5. cardiac function was normal, left ventricular ejection fraction (LVEF) ≥ 50% detected by two-dimensional echocardiography.
* Fertile male or female patients voluntarily used effective contraceptive methods during the study period and within 6 months of the last study, such as double barrier contraceptives, condoms, oral or injection contraceptives, intrauterine devices, etc. All female patients will be considered fertile unless the female patient has undergone natural menopause, artificial menopause or sterilization (such as hysterectomy, bilateral adnexectomy or radioactive ovarian irradiation).
* Puncture biopsy to determine tumor pathology type as ICC.

Exclusion Criteria:

* Participated in clinical trials of other antineoplastic drugs within 4 weeks before entering the group.
* Received any surgery or invasive treatment or operation (except venous catheterization, puncture and drainage, etc.) within 4 weeks before the start of the group;
* History of hepatectomy, history of TACE treatment, previous immune and targeted therapy;
* gene sequencing identified alterations in FGFR2, such as fusions or rearrangements；
* The researchers determined that liver metastases accounted for 70% or more of the total liver volume;
* Patients who have previously received organ transplants or planned organ transplants;
* Patients with obstructive jaundice but not as expected;
* Suffered from other malignant tumors in the past 5 years, except basal cell or squamous cell carcinoma of the skin after radical resection, or cervical carcinoma in situ;
* Patients who have had any brain metastases or are currently suffering from brain metastases;
* In the first study, he took other strong inducers or inhibitors of CYP3A4 within 2 weeks before medication;
* Received any operation (except biopsy) or invasive treatment or operation within 4 weeks before the start of the group, and the surgical incision did not completely heal (except venous catheterization, puncture and drainage, etc.);
* The researchers judged clinically significant electrolyte abnormalities;
* At present, the patients have hypertension that cannot be controlled by drugs, which is defined as systolic blood pressure ≥ 140 mmHg and / or diastolic blood pressure ≥ 90 mmHg.
* Urine routine showed that the amount of urinary protein was more than 2 grams and the amount of 24-hour urinary protein was more than 1.0 g.
* The researchers determined that during the follow-up study, the tumor was most likely to invade important blood vessels and cause fatal massive bleeding;
* Patients with obvious evidence or history of bleeding tendency within 3 months (bleeding > 30 mL within 3 months, hematemesis, black feces, hematochezia), hemoptysis (fresh blood > 5 mL within 4 weeks), hereditary or acquired history of bleeding or coagulation dysfunction. There were significant clinical bleeding symptoms or definite bleeding tendency in the first 3 months, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, etc.;
* Cardiovascular diseases with significant clinical significance, including, but not limited to, acute myocardial infarction, severe / unstable angina pectoris or coronary artery bypass grafting within 6 months before admission; congestive heart failure New York Heart Association (NYHA) grade > 2; ventricular arrhythmias requiring medication; electrocardiogram (ECG) showed QTc interval ≥ 480ms;
* Active or uncontrolled severe infection (≥ （Common Terminology Criteria for Adverse Events）CTCAE 2 grade infection);
* Due to any unalleviated toxicity higher than CTCAE 1 grade caused by any previous anticancer therapy, excluding alopecia, lymphocytopenia and oxaliplatin-induced neurotoxicity ≤ 2;
* Women who are pregnant (positive for pre-medication pregnancy test) or breastfeeding;
* Any other disease, with clinically significant metabolic abnormalities, physical examination abnormalities or laboratory abnormalities, according to the researchers, there is reason to suspect that the patient has a disease or state that is not suitable for the use of research drugs (such as having seizures and requiring treatment), or will affect the interpretation of the results of the study, or put the patient at high risk;
* Known human immunodeficiency virus (HIV) infection
* Patients with any active, known or suspected autoimmune diseases (including but not limited to: myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, enteritis, multiple sclerosis, vasculitis, glomerulonephritis, uveitis, hypophysitis, hyperthyroidism, etc.)
* Known to have allergic reactions to other monoclonal antibodies or to any component of sovantinib;
* The researchers judged that patients have other factors that may affect the results of the study or lead to the termination of the study, such as alcohol abuse, drug abuse, and other serious diseases (including mental illness) that need to be combined with treatment. there are serious laboratory abnormalities, accompanied by family or social factors, which will affect the safety of patients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Objective remission rate (ORR) | After the first DEB-TACE treatment, until the disease progresses or dies (during the treatment of the patient) or the toxicity is intolerable，through study completion, an average of 1 year
  Refers to the proportion of patients whose tumors have shrunk to a certain amount and maintained for a certain period of time, including cases of complete remission (CR), partial remission (PR).

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Refers to the date from the date of admission to the date of the first progression of disease or death of any cause.
Disease control rate (DCR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
  Percentage of confirmed cases including complete remission (CR), partial remission (PR) and disease stability (SD) among patients with evaluable efficacy
Total Survival time (OS) | Through study completion, an average of 1 year
  Refers to the date from the date of admission to the date of death of any cause
Incidence of adverse events and toxicities of Surufatinib in combination with Camrelizumab | Until the last medication for 30 days (±7 days) or before the start of other anti-tumor therapy (whichever occurs first).
  Categorized according to NCI Common Toxicity Criteria version 5.0. Summarized in terms of type, severity (grade 1-5), and dose level in tabular format.

CONTACTS AND LOCATIONS:
Overall Officials: Wanguang Zhang, M.D.,Ph.D., Principal Investigator — Medical Ethics Committee of Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Derived] Guo B, Fan Y, Li D, Xia F, Luo C, Zhu J, Wu Y, Zhu Z, Xiang S, Liu E, Zhang W. Locoregional gemcitabine plus surufatinib and camrelizumab in FGFR2-non-altered intrahepatic cholangiocarcinoma. Cell Rep Med. 2025 Dec 16;6(12):102482. doi: 10.1016/j.xcrm.2025.102482. Epub 2025 Dec 4. PMID 41349529